CLINICAL TRIAL: NCT05096052
Title: PROlectin M, a Nucleocapsid TErminal GaleCTin Antagonist for COVID-19 (PROTECT), a Randomized, Double-blinded, Placebo-controlled Clinical Trial to Evaluate the Efficacy and Safety Among Asymptomatic to Moderately-severe, Ambulatory Patients.
Brief Title: PROlectin M, a Nucleocapsid TErminal GaleCTin Antagonist for COVID-19
Acronym: PROTECT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bioxytran Inc. (Industry)
Collaborators: ALKE RESEARCH PRIVATE LIMITED (Unknown); Research Consultancy (Unknown)
Responsible Party: Principal Investigator, DR ALBEN SIGAMANI, Consultant MD Physician, Bioxytran Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALKE20001
Record Dates: First submitted 2021-10-21; First posted 2021-10-27 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: COVID-19; COVID-19 Pandemic; COVID-19 Respiratory Infection; SARS-CoV2 Infection; Cytokine Release Syndrome
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome | interventions — galactomannan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ProLectin M (Experimental): Active chewable tablets containing galectin inhibitor complex carbohydrate
  Interventions: Drug: Galactomannan
- PLACEBO (Placebo Comparator): Placebo chewable tablets not containing galectin inhibitor complex carbohydrate
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: Galactomannan — Precise chemistry based molecule that binds to galectin like receptors on the N terminal of S1 subunit of the Sars-CoV2 virus
  Arms: ProLectin M
Drug: PLACEBO — A blinded matching placebo containing inert chemistry not able to recognise and bind to the galectin like receptors on the N terminal of S1 subunit of the Sars-CoV2 virus
  Arms: PLACEBO

SUMMARY:
A galectin antagonist prevents viral entry of Sars-CoV-2 virus by blocking the specific terminal on the surface receptors that enables the virus to enter human cells. This inhibitor - ProLectin M is a novel substance that is given orally to individuals who have an infection with Sars-CoV-2 or its subsequent mutations causing COVID19 disease. The oral tablet is chewed every hour, for 8 hours daily, for 7 days.

We hypothesize that patients receiving the active investigational product (ProLectin M), irrespective of their vaccination status, or underlying medical conditions, will have a faster recovery from COVID19 compared to those receiving its matching placebo. The trial is approved by an Institutional Review Board for safety and all participants will need to provide written informed consent to participate in this trial. The safety of ProLectin M is established as the drug substance is recognised as a safe substance. However, its benefits in relieving patients from the COVID19 infection and providing the patients faster recovery from its clinical symptoms and prevention of delayed sequelae of the infection has not been proven yet.

DETAILED DESCRIPTION:
SarsCov2 causes inflammation by releasing cytokines. This is caused by the expressed galectins which are immunogenic.

Binding of the virus to human galectins also give it a very unique property to stealthily avoid the human innate immune system. This is the reason why even present day vaccines are failing to prevent spread of infections.

In this background, our investigational drug has the unique ability to mimic human Galectin 3 and prevent viral entry into host cells. This makes the virus vulnerable to our natural innate immune system to clear it from the oro pharyngeal and GITract.

Randomizing patients into active and placebo groups in a blinded placebo controlled trial can provide us evidence on the ability of ProLectin M to eliminate the virus and prevent even spread of the virus in the community. This also will demonstrate for the first time, how carbohydrates can be used to block significantly infection causing viruses in human beings.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female patient of ≥ 18 years of age, regardless of vaccine status or viral variant or underlying medical conditions, willing and able to provide written informed consent for participation in the study and ready to comply with the study procedures and schedule.
2. Patient having a positive diagnosis for the presence of SARS-CoV-2, obtained from a recently performed rRT-PCR (≤ 3 days) with any 1 of the following:

   i. Ct value ≤ 25 ii. Hospitalized for having classical (CDC defined) symptoms of COVID-19 (onset ≤ 5 days) iii. High risk category of COVID-19: blood group type A-positive type 2 diabetes, or other chronic disease known to have higher morbidity risk with SARS-CoV-2 infection.
3. Patient has the ability to take oral medication and be willing to adhere to the trial protocol regimen of repeated swab collections and frequent follow up for 29 days.
4. Females of child bearing potential who has been using a highly effective contraception for at least 1 month prior to screening and agrees to continue using it during the study participation/enrolment, confirmed through negative pregnancy test

Exclusion Criteria:

* 5. Oxygen Saturation levels (SpO2) ≤ 94% on room air. 6. Female patients who are pregnant or breastfeeding. 7. Patients with any active malignancy or undergoing active chemotherapy. 8. Patients who are currently receiving or have received any investigational treatment for COVID-19 within 30 days prior to screening.

  9. In the opinion of the Investigator, the participation of the patient in the study is not in the patient's best interest, or the patient has any medical condition that does not allow the study protocol to be followed safely.

  10. Patients with known allergies to any of the components used in the formulation of the interventions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-09-25 (Estimated)

PRIMARY OUTCOMES:
Change in seropositivity from baseline for-detection of viral shedding | 14 days
  detecting quantitative SARS-CoV-2 in nasopharynx at intervals of days 1,2, 3, 5, 7, 9 and 14
Change in clinical status from baseline | 14 days
  Proportion of patients reporting improvement in their disease on a WHO Clinical Progression Scale measured daily over the course of the study

SECONDARY OUTCOMES:
time to discharge or to a NEWS of ≤ 2 | 29 days
Duration of hospitalisation | 29 Days
mortality / Serious adverse events | 29 Days

IPD SHARING:
Plan to Share IPD: Undecided
The sponsors and the study representatives and other stakeholders will take a decision on completion of the trial